CLINICAL TRIAL: NCT00824434
Title: A Prospective, Multi-center Trial to Assess an Everolimus-Eluting Coronary Stent System (PROMUS Element™)
Acronym: PLATINUM QCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2051
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: Atherosclerosis; Coronary Artery Disease
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Stent (Experimental)
  Interventions: Device: PROMUS Element™

INTERVENTIONS:
Device: PROMUS Element™ — Drug eluting coronary stent system

SUMMARY:
Compile acute (30-day) clinical outcomes data and 9-month angiographic and intravascular ultrasound (IVUS) data for the PROMUS Element™ Everolimus- Eluting Coronary Stent System in the treatment of patients with a single de novo atherosclerotic lesion

ELIGIBILITY:
Inclusion Criteria:

* Patient (or legal guardian) understands the study requirements and the treatment procedures and provides written informed consent before any study-specific tests or procedures are performed
* Patient is eligible for percutaneous coronary intervention (PCI)
* Patient has documented stable angina pectoris (Canadian Cardiovascular Society [CCS] Classification 1, 2, 3, or 4) or documented silent ischemia; or unstable angina pectoris (Braunwald Class IB-C, IIB-C, or IIIB-C)
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG)
* Patient has a left ventricular ejection fraction (LVEF) >=30% as measured within 30 days prior to enrollment
* Patient is willing to comply with all specified follow-up evaluations

Angiographic Inclusion Criteria:

* Target lesion must be a de novo lesion located in a native coronary artery with visually estimated diameter of >=2.25 mm and <=4.25 mm
* Target lesion length must measure (by visual estimate) <=34 mm
* Target lesion must be in a major coronary artery or branch with visually estimated stenosis >=50% and <100% with Thrombolysis in Myocardial Infarction (TIMI) flow >1.

Exclusion Criteria:

* Patient has clinical symptoms and/or electrocardiogram (ECG) changes consistent with acute myocardial infarction (MI)
* Patient has had a known diagnosis of recent MI (within 30 days prior to the index procedure) and has elevated enzymes at the time of the index procedure as follows.

  * Patients are excluded if any of the following criteria are met at the time of the index procedure

    * If creatine kinase, MB band (CK-MB) >2× upper limit of normal (ULN), the patient is excluded regardless of the creatine kinase (CK) Total.
    * If CK-MB is 1-2× ULN, the patient is excluded if the CK Total is >2× ULN.
  * If CK Total/CK-MB are not used and Troponin is, the patients are excluded if the following criterion is met at the time of the index procedure.

    * Troponin >1× ULN with at least one of the following.

      * Patient has ischemic symptoms and electrocardiogram (ECG) changes indicative of ongoing ischemia (e.g., >1mm ST segment elevation or depression in consecutive leads or new left bundle branch block [LBBB]);
      * Development of pathological Q-waves in the ECG
      * Imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.

Note: For patients who have had a recent MI, CK Total/CK-MB (or Troponin if CK Total/CK-MB are not used) must be documented prior to enrolling the patient

* Patient has received an organ transplant or is on a waiting list for an organ
* transplant
* Patient is receiving or scheduled to receive chemotherapy within 30 days before or after the index procedure
* Patient is receiving oral or intravenous immunosuppressive therapy (ie, inhaled steroids are not excluded) or has known life-limiting immunosuppressive or autoimmune disease (e.g., human immunodeficiency virus, systemic lupus erythematosus, but not including diabetes mellitus)
* Patient is receiving chronic (>=72 hours) anticoagulation therapy (eg, heparin, coumadin) for indications other than acute coronary syndrome
* Patient has a platelet count <100,000 cells/mm3 or >700,000 cells/mm3
* Patient has a white blood cell (WBC) count <3,000 cells/mm3
* Patient has documented or suspected liver disease, including laboratory evidence of hepatitis
* Patient is on dialysis or has known renal insufficiency (i.e., estimated creatinine clearance <50 mL/min by the Cockcroft Gault formula, ie [(140-age)*lean body weight (in kg)]/[plasma creatinine (mg/dL)*72])
* Patient has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Patient has had a cerebrovascular accident (CVA) or transient ischemic attack (TIA) within the past 6 months, or has any permanent neurologic defect that may cause non-compliance with the protocol
* Target vessel or side branch has been treated with any type of percutaneous coronary intervention (PCI; eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 12 months prior to the index procedure
* Target vessel has been treated within 10 mm proximal or distal to the target lesion (by visual estimate) with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) at any time prior to the index procedure
* Non-target vessel or side branch has been treated with any type of PCI (eg, balloon angioplasty, stent, cutting balloon, atherectomy) within 24 hours prior to the index procedure
* Planned or actual target vessel treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon or transluminal extraction catheter immediately prior to stent placement
* Planned percutaneous coronary intervention or coronary artery bypass grafting after the index procedure
* Patient previously treated at any time with coronary intravascular brachytherapy
* Patient has a known allergy to the study stent system or protocol-required concomitant medications (e.g., stainless steel, platinum, cobalt, chromium, nickel, tungsten, acrylic, fluoropolymers, everolimus, thienopyridines, aspirin, contrast) that cannot be adequately premedicated
* Patient has active peptic ulcer or active gastrointestinal (GI) bleeding
* Patient has one of the following:

  * Other serious medical illness (eg, cancer, congestive heart failure) that may reduce life expectancy to less than 24 months
  * Current problems with substance abuse (eg, alcohol, cocaine, heroin, etc.)
  * Planned procedure that may cause non-compliance with the protocol or confound data interpretation
* Patient is participating in another investigational drug or device clinical trial that has not reached its primary endpoint
* Patient intends to participate in another investigational drug or device clinical trial within 12 months after the index procedure
* Known intention to procreate within 12 months after the index procedure
* Female with positive pregnancy test within 7 days prior to the index procedure (a pregnancy test must be performed in women of child-bearing potential prior to enrollment), or lactating
* Patient has more than 1 target lesion or more than 1 target lesion and 1 non-target lesion, identified during screening for intervention

Angiographic Exclusion Criteria:

* Target lesion meets any of the following criteria:

  * Aorto-ostial location (i.e., lesion located within 5 mm of the ostium)
  * Left main location
  * Located within 5 mm of the origin of the left anterior descending (LAD) coronary artery or left circumflex (LCX) coronary artery
  * Located within a saphenous vein graft or an arterial graft
  * Can only be accessed via a saphenous vein graft or an arterial graft
  * Involves a side branch >=2.0 mm in diameter
  * Involves a clinically significant side branch <2.0 mm in diameter that has a clinically significant stenosis at the ostium
  * TIMI flow 0 (total occlusion) or TIMI flow 1 prior to wire crossing
  * Excessive tortuosity proximal to or within the lesion
  * Extreme angulation proximal to or within the lesion
  * Target lesion and/or target vessel proximal to the target lesion is moderately to severely calcified
  * Restenotic from previous intervention
  * Thrombus, or possible thrombus, present in the target vessel
* Patient has an additional clinically significant lesion(s) in the target vessel for which an intervention within 12 months after the index procedure is likely to be required

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian T. Meredith, MBBS, Principal Investigator — Monash Medical Centre
Locations (17):
- Australia (9):
  - St. Vincent's Hospital - Sydney, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Monash Medical Centre, Clayton, Victoria
  - St. Vincent Hospital (Melbourne), Fitzroy, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - Royal Adelaide Hospital, Adelaide
  - The Prince Charles Hospital, Brisbane
  - Liverpool Hospital, Liverpool
  - Sir Charles Gairdner Hospital, Perth
- Institut Jantung Negara, Kuala Lumpur, Malaysia
- New Zealand (5):
  - Middlemore Hospital, Otahuhu, Auckland
  - North Shore Hospital, Takapuna, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Wellington Hospital, Wellington
- Singapore (2):
  - National University Hospital, Singapore, Singapore, Singapore
  - National Heart Centre Singapore, Singapore, Singapore

REFERENCES:
- [Result] Meredith IT, Whitbourn R, Scott D, El-Jack S, Zambahari R, Stone GW, Teirstein PS, Starzyk RM, Allocco DJ, Dawkins KD. PLATINUM QCA: a prospective, multicentre study assessing clinical, angiographic, and intravascular ultrasound outcomes with the novel platinum chromium thin-strut PROMUS Element everolimus-eluting stent in de novo coronary stenoses. EuroIntervention. 2011 May;7(1):84-90. doi: 10.4244/EIJV7I1A15. PMID 21550907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment of 100 subjects was planned, 100 were enrolled at 14 investigative sites in the Asia Pacific region by July 22, 2009.
Groups:
- PROMUS Element: Participants who were treated with the PROMUS Element everolimus-eluting stent (investigational device)
Period: Overall Study
Arm/Group | PROMUS Element
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 60
  >=65 years | 40
Age Continuous [Mean (Standard Deviation); unit: years] | 61.82 (9.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 77
Race/Ethnicity, Customized [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Asian | 16
    Caucasian | 78
    Maori | 1
    Native Hawaiian or other Pacific Islander | 2
    Other | 3
Region of Enrollment [Number; unit: participants]
  Malaysia | 9
  Singapore | 3
  Australia | 49
  New Zealand | 39
General Medical History [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Smoking, Ever | 64
    Medically Treated Diabetes | 19
    Hyperlipidemia Requiring Medication | 81
    Hypertension Requiring. Medication | 66
    History of Bleeding Disorder | 3
Cardiac History [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    Stable Angina | 57
    Unstable Angina | 38
    No Angina | 5
    Silent Ischemia | 2
    Family History of Coronary Artery Disease | 49
    Previous MI | 39
    History of Percutaneous Coronary Intervention | 31
    History of Coronary Artery Bypass Graft | 5
    History of Arrhythmia | 4
    History of Multivessel Disease | 34
    History of Left Main Disease | 2
Cardiac History-Left Ventricular Ejection Fraction [Mean (Standard Deviation); unit: Percent ejection fraction] | 64.41 (13.30)
Neurologic History [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    History of Transient Ischemic Attack | 2
    History of Cerebrovascular Accident | 3
Renal and Peripheral History [Number; unit: Participant] — The same participant may be included in more than one category therefore the number of participants for this baseline measure does not equal the total number of participants in the group.
  Participant
    History of Renal Disease | 1
    History of Peripheral Vascular Disease | 3
Lesion Characteristic-Target Vessel [Number; unit: Lesion]
  Left Anterior Descending Artery | 35
  Left Circumflex Artery | 30
  Right Coronary Artery | 35
Lesion Location [Number; unit: Lesions]
  Proximal | 37
  Mid | 54
  Distal | 7
  Ostial | 2
Lesion Characteristics [Mean (Standard Deviation); unit: millimeters]
  Reference Vessel Diameter | 2.72 (0.53)
  Minimum Lumen Diameter | 0.71 (0.34)
  Lesion Length | 15.40 (7.03)
Lesion Characteristic-Diameter Stenosis [Mean (Standard Deviation); unit: Percent Diameter Stenosis] | 74.09 (10.93)
Lesion Characteristics [Number; unit: Lesions] — The same lesion may be included in more than one category therefore the number of lesions for this baseline measure does not equal the total number of lesions or participants in the group.
  Lesions
    Eccentric Lesion | 53
    Bend >45% | 12
    Tortuosity | 9
    Calcification, any | 18
    Total Occlusion | 1
    Branch Vessel Disease | 6
Lesion Characteristics: American College of Cardiology (ACC)/American Heart Association (AHA) Class [Number; unit: Lesions] — Type A lesions: minimally complex, readily accessible, non-angulated, smooth contour, little to no calcification, less than totally occlusive, not ostial in location, no major side branch involvement, and an absence of thrombus.
  Type B lesions: moderately complex, eccentric, moderate tortuosity and angulation, moderate or heavy calcification, total occlusion < 3 months old, ostial in location, with presence of thrombus.
  Type C lesions: severely complex, diffuse, excessive tortuosity and angulation, total occlusions > 3 months old, degenerated vein grafts and friable lesions.
  Lesions
    A | 5
    B1 | 28
    B2 | 42
    C | 25
Pre-Procedure Thrombolysis In Myocardial Infarction (TIMI) Flow [Number; unit: Lesion] — TIMI 0 - No perfusion TIMI 1 - Penetration with minimal perfusion TIMI 2 - Partial perfusion TIMI 3 - Complete perfusion
  Lesion
    0 | 1
    1 | 0
    2 | 1
    3 | 98

OUTCOME MEASURES:

1. Primary Outcome: Cardiac Events (Composite)
Description: Percentage of patients who had a myocardial infarction, cardiac death, target lesion revascularization, or stent thrombosis (defined as definite or probable per the Academic Research Consortium [ARC] definitions); see below for definitions of individual components.
Time Frame: 30 days
Population: Analysis was intention to treat; all patients in the study underwent clinical follow up to provide the information needed for this endpoint.
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

2. Secondary Outcome: In-stent Late Loss
Description: In-stent late loss by quantitative coronary angiography in workhorse target lesions (visual reference vessel diameter [RVD] ≥2.5 mm and ≤4.25 mm and visual lesion length ≤24 mm)
Time Frame: 9 months
Population: Analysis was intention to treat; all patients in the study with workhorse lesions (visual reference vessel diameter [RVD] ≥2.5 mm and ≤4.25 mm and visual lesion length ≤24 mm) underwent clinical follow up to provide the information needed for this endpoint.
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | PROMUS Element
Number analyzed (Participants) | 73
millimeters | 0.17 (0.25)
Statistical Analysis 1: Comparison: PROMUS Element; The Student t-test was used to compare the outcome to a prespecified performance goal of 0.44 mm based on an historical TAXUS Express workhorse 9-month in-stent late loss (0.41 mm) value plus delta (0.03 mm); Test type: Superiority or Other; p < 0.0001, t-test, 1 sided; Mean In-stent Late Loss in WH Lesions = 0.17, 95% CI 1-sided [upper limit 0.22]

3. Secondary Outcome: Occurance of Post-procedure Incomplete Stent Apposition
Description: Percentage of participants who experience incomplete stent apposition as determined immediately post-procedure by intravascular ultrasound
Time Frame: Post-procedure
Population: Participants who were treated with the PROMUS Element everolimus-eluting stent (investigational device) and who underwent intravascular ultrasound to determine extent of stent apposition
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 88
percentage of participants | 5.7
Statistical Analysis 1: Comparison: PROMUS Element; A one-sided 95% Clopper-Pearson upper confidence bound was derived and tested to determine if the outcome was less than a prespecified performance goal based on historical XIENCE V/PROMUS post-procedure incomplete apposition data from the SPIRIT III study (34.4%); Test type: Superiority or Other; p < 0.0001, One-sided exact binomial test; Percent Post-procedure Incomplete Apposi = 5.7, 95% CI 1-sided [upper limit 11.6]

4. Secondary Outcome: Myocardial Infarction (MI)
Description: New Q-waves in ≥2 leads lasting ≥0.04 sec with creatine kinase myoglobin band(CK-MB) or troponin >upper limit of normal(ULN); if no new Q-waves total CK levels >3×ULN (peri-percutaneous coronary intervention [PCI]) or >2×ULN (spontaneous) with elevated CK-MB or troponin >3×ULN (peri-PCI) or >2×ULN (spontaneous) plus ≥one of the following: ECG changes indicating new ischemia (new ST-T changes, left bundle branch block), imaging evidence of new loss of viable myocardium, new regional wall motion abnormality. Similar for MI diagnosis post coronary artery bypass graft with CK-MB or troponin >5×ULN
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 0.0

5. Secondary Outcome: All-cause Mortality
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 0.0

6. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: Target lesion revascularization (TLR) is any ischemia-driven repeat percutaneous intervention to improve blood flow of the successfully treated target lesion or bypass surgery of the target vessel with a graft distally to the successfully treated target lesion.
Time Frame: 30 Days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

7. Secondary Outcome: Target Lesion Revascularization (TLR)
Description: as for outcome 6
Time Frame: 12 Months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

8. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: Target vessel revascularization (TVR) is any ischemia-driven repeat percutaneous intervention to improve blood flow, or bypass surgery of not previously existing lesions with diameter stenosis ≥50% by quantitative coronary angiography in the target vessel, including the target lesion.
Time Frame: 30 Days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

9. Secondary Outcome: Target Vessel Revascularization (TVR)
Description: as for outcome 8
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

10. Secondary Outcome: Target Lesion Failure (TLF)
Description: Target lesion failure (TLF) is defined as any ischemia-driven revascularization of the target lesion, myocardial infarction (Q-wave and non-Q-wave) related to the target vessel, or cardiac death related to the target vessel.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

11. Secondary Outcome: Target Vessel Failure (TVF)
Description: Target vessel failure (TVF) is defined as any ischemia-driven revascularization of the target vessel, myocardial infarction (MI, Q-wave and non-Q-wave) related to the target vessel or death related to the target vessel. For the purposes of this protocol, if it cannot be determined with certainty whether the MI or death was related to the target vessel, it will be considered a TVF.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

12. Secondary Outcome: Definite + Probable Stent Thrombosis Based on Academic Research Consortium (ARC) Definition
Description: DEFINITE ST: acute coronary syndrome and angiographic or pathologic evidence of stent thrombosis; PROBABLE ST: unexplained death within 30 days or target-vessel infarction without angiographic information ARC ST is reported as a cumulative value at different time points and within the different separate time points. Time 0 is the time point after the guide catheter has been removed. Acute ST: 0-24 hours after stent implantation; Subacute ST: >24 hours to 30 days post; late ST: >30 days to 1 year post; Very late ST: >1 year post; NOTE: Acute/subacute can be replaced by early ST (0-30 days).
Time Frame: 24 hours
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 1.0

13. Secondary Outcome: Definite + Probable Stent Thrombosis Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 12
Time Frame: >24 hr-30 days
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 0.0

14. Secondary Outcome: Definite + Probable Stent Thrombosis Based on Academic Research Consortium (ARC) Definition
Description: as for outcome 12
Time Frame: >30 days-1 year
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 0.0

15. Secondary Outcome: Clinical Procedural Success
Description: Mean lesion diameter stenosis < 30% with TIMI 3 flow without the occurrence of in-hospital cardiac death, MI, or TVR
Time Frame: Duration of hospital stay (usually 1-2 days)
Population: Analysis was intention to treat
Measure: Number; unit: percentage of participants
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
percentage of participants | 99.0

16. Secondary Outcome: Technical Success
Description: Successful delivery and deployment of the study stent to the target lesion, without balloon rupture or embolization, summarized per stent.
Time Frame: Acute-At time of index procedure
Population: Intention to treat
Measure: Number; unit: percentage of stents attempted
Units Other Than Participants: stents attempted in the target vessel
Arm/Group | PROMUS Element
Number analyzed (Participants) | 100
Number analyzed (stents attempted in the target vessel) | 108
percentage of stents attempted | 100.0

ADVERSE EVENTS:
Time Frame: Site reported adverse events were collected through 365 days.
Arm/Group | PROMUS Element
Serious Adverse Events (participants affected / at risk) | 27/100
Other Adverse Events (participants affected / at risk) | 48/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=100)
Angina pectoris (Cardiac disorders) | 4 (5)
Angina unstable (Cardiac disorders) | 3 (5)
Coronary artery dissection (Cardiac disorders) | 3 (4)
Myocardial infarction (Cardiac disorders) | 2 (2)
Arteriospasm coronary (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Coronary artery thrombosis (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 8 (8)
Catheter site discharge (General disorders) | 1 (1)
Catheter site haemorrhage (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1)
Macular hole (Eye disorders) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Intermittant claudication (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PROMUS Element (N=100)
Non-cardiac chest pain (General disorders) | 8 (9)
Angina pectoris (Cardiac disorders) | 7 (7)
Catheter site haematoma (General disorders) | 7 (8)
Adverse drug reaction (General disorders) | 6 (7)
Catheter site discharge (General disorders) | 6 (7)
Chest pain (General disorders) | 5 (5)
Coronary artery dissection (Cardiac disorders) | 8 (8)
Myocardial infarction (Cardiac disorders) | 8 (8)
Troponin increased (Investigations) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator shall have the right to publish the results, provided that before publishing, the PI shall submit copies of any proposed publication or presentation to Sponsor for review at least 40 days in advance of submission for publication or presentation to a publisher or other third party. Sponsor reserves the right to delete any confidential information or other proprietary information of Sponsor from the proposed publication or presentation.